CLINICAL TRIAL: NCT02422628
Title: Correlation Between Epithelial Growth Factor Receptor(EGFR) Mutation Using cfDNA and CTCs in Patients With Non-Small Cell Lung Cancer
Brief Title: Correlation Between EGFR Mutation Using cfDNAs and Circulating Tumor Cells in Patients With NSCLC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201304074RIPC
Record Dates: First submitted 2015-03-29; First posted 2015-04-21 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: EGFR inhibitor; EGFR mutation; EGFR; adenocarcinoma; EGFR TKI; treatment; Non small cell
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples every 3 months till disease progression or intolerable due to side effect.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- EGFR mutation postive: Blood samples every 3 months till disease progression or intolerable due to side effect.
- EGFR mutation wild type: Blood samples before treatment once.
- Healthy Volunteers: Blood samples once.

SUMMARY:
Correlation of epithelial growth factor receptor mutation in blood of lung cancer patient and clinical outcome.

DETAILED DESCRIPTION:
EGFR tyrosine kinase mutation is frequently seen in our NSCLC, especially adenocarcinoma.1 The epidermal growth factor receptor (EGFR) of receptor tyrosine kinases (TKs) regulate many developmental, metabolic and physiological processes. In tumor cells, the TK activity of EGFR may be dysregulated by several mechanisms, including EGFR gene mutation, increased gene copy number and EGFR protein overexpression.1 Improper activation of EGFR TK results in increased malignant cell survival, proliferation, invasion and metastasis. EGFR overexpression is observed in tumors from more than 60% of patients with metastatic non-small-cell lung cancer (NSCLC) and is correlated with poor prognosis.2 Treatment with the reversible EGFR TK inhibitors (TKIs), gefitinib and erlotinib, results in dramatic antitumor activity in a subset of patients with NSCLC. Sequencing of the EGFR gene revealed that a majority of tumors responding to EGFR TKIs harbored mutations in the TK domain of EGFR. For patients whose tumors exhibit EGFR mutations, the response rate to gefitinib and erlotinib is approximately 75%, suggesting that these mutations, at least in part, drive malignant transformation.

However, the disease-free time to progression was still less than 1 year in most study.3-5 More than half of patients acquired resistant by new EGFR T790M resistance mutation. A second biopsy at the time of progression is becoming an issue. However, Only around 30% of NSCLC patients can receive gene testing to predict target therapy response because of the risk and difficulty in obtaining adequate tissues from the primary lung tumors by biopsy. Serial monitoring the emergence of resistant mutations is almost not possible. Recently, circulating free DNAs (cfDNAs) become a promising topic in cancer research. cfDNA can be used as a liquid biopsy, allowing repeated blood samples to be taken and changes in mutation status to be tracked throughout a cancer treatment, paving the way for a potential use in following up of treatment response, gauging prognosis, or monitoring of recurrence.6 It has been known for over a hundred years that disseminated tumor cells can be found in the circulation of patients with metastatic cancer and it has been hypothesized that these circulating tumor cells (CTCs) may represent cancer stem cells or a high metastatic potential cellular population.7 The major challenge since as few as one CTC may be found in the background of 105-106 peripheral blood mononuclear cells.8 CTCs are an attractive alternative to tumor tissue for biomarker analysis including EGFR mutation. CTCs can be obtained from a routine blood draw with minimal risk and inconvenience to the patient compared to a fresh biopsy. Another appealing facet of CTCs as a surrogate diagnostic tissue is the idea that CTCs could also constitute a "liquid biopsy" like cfDNA and provide real-time information about the patient's current disease state.9,10 Analysis of biomarker status in CTCs collected prior to treatment could potentially be used to select an appropriate targeted therapy, while repeated longitudinal sampling during treatment could be used to detect appearance of resistance markers and potentially enable switching to a more appropriate therapy.

A side-by-side comparison of EGFR mutation analysis in DNA extracted from circulating tumour cells (CTCs) versus cfDNA from plasma suggested that mutational analysis of CTCs captured on the CellSearch platform was low by comparison with the frequency of EGFR mutations identified in plasma.11 However, this limitation might be related to the CellSearch platform used,11 because other CTC platforms (eg, CTC biochip) have greater sensitivity and specificity for EGFR mutational analyses.12 New technologies, such as next generation sequencing and digital PCR (Figure 1), which can permit more precise quantification of cfDNA and also the CTCs, offer opportunities to design more appropriate treatments. Longitudinal analyses of EGFR and other mutations in cfDNA and CTCs might well prove to be an ideal non-invasive technique to be included in the oncologist's repertoire at the time of assigning or monitoring treatment in patients with NSCLC.

In this study, the investigators will collect blood from NSCLC patients who harbor EGFR mutation in biopsy specimens. Buffy coat and serum/plasma will be separated and DNA will be extracted. The investigators will check the EGFR mutation by next generation sequencing or digital PCR. Blood from volunteers without lung cancer patient will be also collected as standard. Serial follow-up the change of EGFR mutation every month in cancer patient will be correlated with clinical course. The Investigators hope the detection of EGFR mutation and serial change in the patient blood could offer as a marker for early diagnosis and early relapse.

ELIGIBILITY:
NSCLC patients should fulfill the following criteria:

1. Provision of informed consent prior to any study specific procedures
2. Patients with non-small cell lung cancer, adenocarcinoma, aged 20 years and older.
3. Tumor harboring EGFR mutation including activating mutation L858R, Del19 or/and resistant mutation T790M, or/and rare mutation G719, S768, L861
4. Treatment naive
5. Patients will receive EGFR-TKI as first line treatment.

For inclusion in the study of control subjects (100 volunteers), they should fulfill the following criteria:

1. Provision of informed consent prior to any study specific procedures
2. Patients aged 20 years and older
3. Volunteers without any lung cancer related diagnosis or symptoms
4. EGFR TKI treatment naïve and without any EGFR TKI treatment in the following process

For inclusion in the study of control subjects (100 EGFR wild-type), they should fulfill the following criteria:

1. Provision of informed consent prior to any study specific procedures
2. Patients with non-small cell lung cancer, adenocarcinoma, aged 20 years and older.
3. Tumor with no EGFR mutation detected (mutation L858R, Del19 or/and resistant mutation T790M, or/and rare mutation G719, S768, L861)
4. EGFR TKI treatment naïve and without any EGFR TKI treatment in the following process

   -------

Exclusion criteria

For exclusion in the study of NSCLC patients and control subjects should fulfill the following criteria:

1. Subjects should not enter the study if any of the following exclusion criteria are fulfilled: Involvement in the planning and/or conduct of the study (applies to staff at the study site)
2. Previous enrolment in the present study
3. As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
4. Evidence of any other significant clinical disorder or laboratory finding that made it undesirable for the patient to participate in the study
5. Pregnancy or breast-feeding

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progressive disease measured by RECIST criteria after receiving 1st line EGFR-TKI | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chi Ho, Principal Investigator — National Taiwan University Hospital No. 7, Chung-Shan South Road, Taipei, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan